CLINICAL TRIAL: NCT06953427
Title: The Impact of Age on Short-term Post-thrombectomy Outcomes in Patients Aged 70 or Beyond With Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Victor C. Kok, MMSc, MD, PhD, FACP, Senior attending staff of the Department of Internal Medicine, Kuang Tien General Hospital
Other Study IDs: KTGH-IN-24-003
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acute Cerebral Ischemia; Endovascular Thrombectomy; Prognosis; Age Factors; Interventional Radiology; Elderly (Aged >70)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute cerebral stroke who underwent endovascular thrombectomy: Only patients who aged 70 or above will be enrolled.

SUMMARY:
A recent Cochrane systematic review of 18 randomized controlled trials (RCTs) comparing endovascular intervention-either mechanical thrombectomy or intra-arterial thrombolysis combined with medical treatment-to conservative medical treatment alone provided high-certainty evidence that endovascular intervention increases the likelihood of achieving a favorable functional outcome (modified Rankin Scale [mRS] score of 0-2) by 50% in patients with acute ischemic stroke (AIS).1 More recently, a cross-Atlantic RCT was conducted to determine whether endovascular therapy (EVT) plus medical care is superior to medical care alone in patients with acute proximal cerebral vessel occlusion in the anterior circulation and large infarcts, regardless of infarct size. The study confirmed a 63% increased odds of a favorable outcome with EVT plus medical care. In real-world registries of EVT for AIS due to large-vessel occlusion in the anterior circulation, approximately one-half of patients are aged 70 and older, while 13% to 39% are aged 80 and beyond. In patients aged 70 and beyond who are EVT-eligible, post-procedure mortality increases progressively with increasing age. A prospective European study found that each additional year of age was associated with an 8% decline in the likelihood of achieving a favorable functional outcome. In elderly patients, increasing age is more than just a number-it reflects a higher likelihood of significant medical comorbidities, polypharmacy, declining functional status, compromised nutritional status, and weakened immune function. Research on age as a predictor of EVT outcomes often compares elderly patients to much younger counterparts. However, contrasting post-EVT outcomes in older adults with those under 70 is neither realistic nor appropriate due to inherent differences in baseline health, comorbidities, and physiological resilience. Therefore, the investigators analyzed a prospectively registered cohort to assess whether age influences post-EVT functional outcomes, using septuagenarians as the control group.

DETAILED DESCRIPTION:
This is a retrospective, single-center cohort study evaluating patients aged ≥70 years with AIS who underwent EVT at Kuang Tien General Hospital, Taichung, Taiwan. A registry has been established by the Department of Interventional Neuroradiology under the supervision by Dr. Pao-Sheng Yen. for patients who The stroke center is nationally accredited for its capability to evaluate and perform EVT for acute ischemic stroke emergencies. The study was approved by the Institutional Review Board (IRB) with an approval certificate numbered KTGH-11415, and informed consent was waived due to the retrospective nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Acute Ischemic Stroke due to large-vessel occlusion (LVO) confirmed by CT angiography or MR angiography
* underwent EVT within the standard treatment window
* available 3-month modified Rankin Scale (mRS) scores.

Exclusion Criteria:

* Premorbid mRS score >2
* Poor imaging quality precluding assessment
* Lack of follow-up data.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Single-center cohort of patients aged ≥70 years with AIS who underwent EVT at Kuang Tien General Hospital, Taichung, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Post-endovascular thrombectomy modified Thrombolysis in Cerebral Infarction (mTICI) reperfusion grade | Immediate post-thrombectomy
  Modified Treatment In Cerebral Ischemia (TICI) scale:
  Score Definition 0: No reperfusion;
  1: Flow beyond occlusion without distal branch reperfusion; 2a: Reperfusion of less than half of the downstream target arterial territory; 2b: Reperfusion of more than half, yet incomplete, in the downstream target arterial territory; 3: Complete reperfusion of the downstream target arterial territory, including distal branches with slow flow.
  This is an immediate post-procedure assessment relating to capillary-level reperfusion as measured on catheter angiography.
Three-months post-EVT modified Rankin scale (mRS) | 3-months post-EVT
  Modified Rankin Scale Score Description 0: No symptoms at all;
  1. No significant disability despite symptoms; able to carry out all usual duties and activities;
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance;
  3. Moderate disability; requiring some help, but able to walk without assistance;
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance;
  5. Severe disability; bedridden, incontinent, and requiring constant nursing care and attention;
  6. Dead.

SECONDARY OUTCOMES:
Spontaneous intracerebral hemorrhage | Day 2 to Day 90 post-EVT
  A CT scan will be performed on day 2 to detect any spontaneous intracerebral hemorrhage. In patients who are fine on day 2, will perform CT scan to check bleeding when symptoms arise.

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Sheng Yen, MD, Study Director — Kuang Tien General Hospital
Locations (1):
- Department of Interventional Neuro-Radiology, Kuang Tien General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Most of the relevant clinical characteristics will be reported as aggregate data.

REFERENCES:
- [Background] 1. Roaldsen MB, Jusufovic M, Berge E, Lindekleiv H. Endovascular thrombectomy and intra-arterial interventions for acute ischaemic stroke. Cochrane Database Syst Rev. 2021 Jun 14;6(6):Cd007574. 2. Costalat V, Jovin TG, Albucher JF, et al. Trial of Thrombectomy for Stroke with a Large Infarct of Unrestricted Size. N Engl J Med. 2024 May 9;390(18):1677-89. 3. Zerna C, Rogers E, Rabi DM, et al. Comparative Effectiveness of Endovascular Treatment for Acute Ischemic Stroke: A Population-Based Analysis. J Am Heart Assoc. 2020 Apr 7;9(7):e014541. 4. Adcock AK, Schwamm LH, Smith EE, et al. Trends in Use, Outcomes, and Disparities in Endovascular Thrombectomy in US Patients With Stroke Aged 80 Years and Older Compared With Younger Patients. JAMA Netw Open. 2022 Jun 1;5(6):e2215869. 5. Enriquez BAB, Halling HK, Lund CG, et al. Exploring the Impact of Age and Pre-Stroke Modified Rankin Scale in Elderly Thrombectomy: A 15-Year Single-Center Experience. Cerebrovasc Dis Extra. 2024;14(1):125-33. 6. Groot AE, Treurniet KM, Jansen IGH, et al. Endovascular treatment in older adults with acute ischemic stroke in the MR CLEAN Registry. Neurology. 2020 Jul 14;95(2):e131-e9. 7. Zhai G, Song J, Yu N, et al. Predictors of Mechanical Thrombectomy for Anterior Circulation Emergent Large-Vessel Occlusion in the Older Adults. Clin Appl Thromb Hemost. 2023 Jan-Dec;29:10760296231184219. 8. Inoue M, Ota T, Hara T, et al. An Initial High National Institutes of Health Stroke Scale Score and Any Intracranial Hemorrhage Are Independent Factors for a Poor Outcome in Nonagenarians Treated with Thrombectomy for Acute Large Vessel Occlusion: The Tokyo/Tama-REgistry of Acute Endovascular Thrombectomy (TREAT) Study. World Neurosurg. 2022 Sep;165:e325-e30. 9. Ippen FM, Schregel K, Ungerer M, Feisst M, Ringleb PA, Gumbinger CK. Outcomes in elderly patients undergoing endovascular thrombectomy in association with premorbid Rankin Scale scores. Front Neurol. 2024;15:1418415. 10. Yen PS, Kok VC, Lin YH, Wu YT,